CLINICAL TRIAL: NCT01648998
Title: The Effects of Fludrocortisone on Information Processing in Healthy Female Volunteers
Brief Title: Fludrocortisone and Information Processing in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Willem Van der Does, Professor, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P12-12
Record Dates: First submitted 2012-05-23; First posted 2012-07-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Depression
Keywords: Mineralocorticoid receptor; Fludrocortisone; Information Processing; Cognition; Depression
MeSH Terms: conditions — Depression | interventions — Fludrocortisone; fludrocortisone acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fludrocortisone (Experimental): Fludrocortisone 500 mg in capsule
  Interventions: Drug: Fludrocortisone
- Placebo (Placebo Comparator): Placebo capsule, single dose, main ingredient lactose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fludrocortisone — single dose 500 mg, capsule
  Other Names: Florinef
  Arms: Fludrocortisone
Drug: Placebo
  Other Names: Placebo comparator
  Arms: Placebo

SUMMARY:
Stimulating the mineralocorticoid receptor (MR) may restore a disturbed balance as seen in depression. In this double-blind, randomized, placebo-controlled trial the investigators will test the effects of a single dose (500mg) fludrocortisone, an MR-agonist, on the information processing in healthy female volunteers (N = 2x20).

The investigators want to investigate whether the acute administration of fludrocortisone (FC) in healthy females enhances the appraisal of emotional information related to depression, hypothesizing that:

* FC relative to placebo selectively improves the recognition of happy and fearful faces: resulting in more correct responses and faster RTs.
* FC induces a bias towards more positive self-description and an improved memory for positive information.

Female participants were selected because the haplotype MRI180V is related to depression vulnerability in women, not in men. If the effects of fludrocortisone are comparable to the effects of antidepressants on the same tests and the same population, it might be a first indication that fludrocortisone may function as an antidepressant.

DETAILED DESCRIPTION:
We found in depressed individuals, compared with non-depressed controls, that MRs had a decreased (approximately -30%) expression in hippocampus, inferior frontal gyrus and cingulate gyrus. It is proposed that decreased expression of MRs is part of the underlying pathological process in depression.

Recent studies have revealed considerable interpersonal differences with regard to the functioning of the MRs. Firstly, common MR gene polymorphisms influence the cortisol awakening response (CAR). Secondly, clinical populations differ in observed depressive symptoms as a function of MRI180V genotype. This MR I180V gene variant showed less activity in vitro, which suggests that functionality in vivo is decreased. Finally, MR haplotype 2, which is prevalent in 35% of the Caucasian population, enhances the transcription, translation and transactivation of the MR. This haplotype is associated with higher dispositional optimism, fewer thoughts of hopelessness and lower risk of major depression. These effects are restricted to pre-menopausal women. This suggests that female sex steroids may interact with the MR gene, thereby modulating resilience. Indeed, it has been shown that progesterone and oestrogen modulate MR-expression in rats. Taken together, mineralocorticoid receptors in the brain are considered to be a new target for the treatment of stress related disorders like depression.

Fludrocortisone (9α fluoro-hydrocortisone) (FC) is a specific MR-agonist currently used to treat diseases of the adrenal cortex, septic shock (Russel, 2008) and occasionally orthostatic hypotension. It is shown that FC significantly inhibits nocturnal HPA axis activity without first depleting MR receptors with an MR-antagonist. This suggests FC have interesting implications in disorders of HPA axis excess, such as depression. Consistent with the idea that the stimulation of the MR might be useful in the treatment of depression, fludrocortisone accelerated the antidepressant effects of the SSRI escitalopram, at least in those patients who responded to escitalopram. This is in line with a previous observation that spironolactone, a MR antagonist, decreased the efficacy of the antidepressant amitriptyline in depressed patients. These studies show that stimulation of the MR might be a useful addition to the treatment of depression. Though, the explanatory mechanism behind these observations remains unclear.

This project is a first step in investigating the potential antidepressant effects of MR stimulation by fludrocortisone. We will test the effects of FC on indices of emotional information processing in healthy volunteers, which is a recently validated model of antidepressant drug action. It has been demonstrated repeatedly that a single dose of an antidepressant changes the processing of emotionally relevant information in healthy volunteers, within a few hours after administration. For instance, one dose of citalopram improved the recognition of facial expressions of fear and happiness relative to placebo in healthy female volunteers. This finding has been replicated with different antidepressants and different populations.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in Dutch
* Age 18-35 yrs
* BMI 18 to 30 kg/m2
* Northwestern European ancestry

Exclusion Criteria:

* Known contra-indications for fludrocortisone use:

  * Allergy to fludrocortisone.
  * Ulcus ventriculi et duodeni.
  * Acute infectious processes; viral infections
  * Tropical worm infections.
  * Vaccination with living virus
* Major physical illness, such as diabetes, thyroid disease, epilepsy, multiple sclerosis, pituitary disease, or any other serious medical condition.
* Hypertension or history of stroke. Increased blood clot formation.
* Major infections.
* Any current or past psychiatric disorder
* Use of medication likely to interfere with the study (e.g., benzodiazepines, St John's Wort).
* Pregnancy or breastfeeding.
* History of regular (more than once per month during three or more months) use of hard drugs (including XTC) or any use during past month.
* Alcohol use of more than 14 units per week or more than 4 units on any day during the week prior to the study or during the study period.
* Regular smoker during past year or use of nicotine product during past week
* Participants will be tested outside their menstrual period (two days before until five days after start of period).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Accuracy to recognize emotions in facial expressions | 2 hrs after intake fludrocortisone or placebo
  This primary outcome is measured by performing the Facial Expression Recognition Task (FERT).
Explicit memory for positive and negative information | 2 hrs after intake of fludrocortisone or placebo
  This primary outcome is measured by the Emotional categorization and Memory(EMT)task. This task consists of two parts, the encoding and recall.

SECONDARY OUTCOMES:
Subjective mood states | 2 hrs after intake fludrocortisone or placebo
  This is measured by administration of the 'Positive Affect Negative Affect Schedule'(PANAS). It measures positive and negative mood states (tension, vigor, anxiety, fatigue, boredom, alertness...) (20 items adding to two subscales, positive and negative affect).

CONTACTS AND LOCATIONS:
Overall Officials: Willem van der Does, Professor, Principal Investigator — Leiden University
Locations (1):
- Leiden University - Institute of Psychology, Leiden, South Holland, Netherlands

REFERENCES:
- [Background] Otte C, Hinkelmann K, Moritz S, Yassouridis A, Jahn H, Wiedemann K, Kellner M. Modulation of the mineralocorticoid receptor as add-on treatment in depression: a randomized, double-blind, placebo-controlled proof-of-concept study. J Psychiatr Res. 2010 Apr;44(6):339-46. doi: 10.1016/j.jpsychires.2009.10.006. Epub 2009 Nov 11. PMID 19909979
- [Background] Klok MD, Vreeburg SA, Penninx BW, Zitman FG, de Kloet ER, DeRijk RH. Common functional mineralocorticoid receptor polymorphisms modulate the cortisol awakening response: Interaction with SSRIs. Psychoneuroendocrinology. 2011 May;36(4):484-94. doi: 10.1016/j.psyneuen.2010.07.024. Epub 2010 Sep 29. PMID 20884124
- [Background] Harmer CJ, Goodwin GM, Cowen PJ. Why do antidepressants take so long to work? A cognitive neuropsychological model of antidepressant drug action. Br J Psychiatry. 2009 Aug;195(2):102-8. doi: 10.1192/bjp.bp.108.051193. PMID 19648538
- [Background] Buckley TM, Mullen BC, Schatzberg AF. The acute effects of a mineralocorticoid receptor (MR) agonist on nocturnal hypothalamic-adrenal-pituitary (HPA) axis activity in healthy controls. Psychoneuroendocrinology. 2007 Sep-Nov;32(8-10):859-64. doi: 10.1016/j.psyneuen.2007.05.016. Epub 2007 Jul 30. PMID 17666187
- [Background] Klok MD, Alt SR, Irurzun Lafitte AJ, Turner JD, Lakke EA, Huitinga I, Muller CP, Zitman FG, de Kloet ER, Derijk RH. Decreased expression of mineralocorticoid receptor mRNA and its splice variants in postmortem brain regions of patients with major depressive disorder. J Psychiatr Res. 2011 Jul;45(7):871-8. doi: 10.1016/j.jpsychires.2010.12.002. Epub 2010 Dec 30. PMID 21195417